CLINICAL TRIAL: NCT02390349
Title: "CuraMed" and "Curamin" in Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EuroPharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EP-1001
Record Dates: First submitted 2015-03-05; First posted 2015-03-17 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- CuraMed (BCM-95) (Experimental): 67 patients, treatment with CuraMed (BCM-95), one capsule (500 mg) orally, three times daily for 12 weeks
  Interventions: Dietary Supplement: CuraMed
- Curamin (Experimental): 67 patients, treatment with Curamin, one capsule (500 mg) orally, three times daily for 12 weeks
  Interventions: Dietary Supplement: Curamin
- Placebo (Placebo Comparator): 67 patients, treatment with placebo, one capsule (500 mg) orally, three times daily for 12 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo
  Arms: Placebo
Dietary Supplement: Curamin
  Arms: Curamin
Dietary Supplement: CuraMed
  Arms: CuraMed (BCM-95)

SUMMARY:
This randomized, placebo-controlled study evaluates the effects of CuraMed ® (BCM-95 ®) and Curamin ® in the treatment of osteoarthritis. One group will receive CuraMed, one group will receive Curamin and one group will receive placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of degenerative hypertrophic osteoarthritis of the knee (M17, according to International Classification of Diseases (ICD-10) of bone joints, verified by radiography (Grade 1-3 by Kellgren-Lawrence radiographic grades).

Exclusion Criteria:

* subjects with inflammatory and any secondary arthritis
* moderate and severe synovitis (grades 2 and 3)
* tear of meniscus
* chronic diseases of the kidneys, liver, gastrointestinal, cardiovascular, endocrine and nervous systems
* allergic anamnesis and drug intolerance
* pregnant or nursing
* history of substance abuse
* subjects taking non-steroidal anti-inflammatory drugs and analgesics within 2 weeks prior to the study
* subjects taking glucosamine sulfate, chondroitin sulfate, intra-articular hyaluronate, systemic or intra-articular glucocorticoids within three months prior to the study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2015-04; Primary Completion 2016-05 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Effect of Curamin and Curamed on joint pain as measured by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 12 weeks
Effects of Curamin and Curamed on physical performance measures using the Osteoarthritis Research Society International (OARSI) tests of physical function | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Erebuni Medical Center, Yerevan, Armenia

REFERENCES:
- [Derived] Haroyan A, Mukuchyan V, Mkrtchyan N, Minasyan N, Gasparyan S, Sargsyan A, Narimanyan M, Hovhannisyan A. Efficacy and safety of curcumin and its combination with boswellic acid in osteoarthritis: a comparative, randomized, double-blind, placebo-controlled study. BMC Complement Altern Med. 2018 Jan 9;18(1):7. doi: 10.1186/s12906-017-2062-z. PMID 29316908